CLINICAL TRIAL: NCT02028351
Title: Comparison of Vision Measured by the Vimetrics Central Vision Analyzer With That Measured by logMAR Acuity Chart Testing Under Similar Conditions of Luminance and Contrast
Brief Title: Vision Measured by the Vimetrics CVA Compared With Chart Testing Under Similar Luminance and Contrast Conditions
Status: Completed | Type: Observational
Sponsor: Sinclair Technologies, LLC (Industry)
Responsible Party: Principal Investigator, Stephen H. Sinclair, MD, Chief Medical Officer, Sinclair Technologies, LLC
Other Study IDs: VVS 001
Record Dates: First submitted 2012-12-29; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Refractive Error; Cataract; Maculopathy
Keywords: visual acuity; contrast sensitivity; cataract; maculopathy
MeSH Terms: conditions — Refractive Errors; Cataract; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal: No Intervention
- Cataract: No intervention
- Maculopathy: No Intervention

SUMMARY:
Purpose of The Study:

The purpose of this study is the following:

A)To gather age-related normative visual acuity data for the Vimetrics Central Vision Analyzer (CVA, Vimetrics, LLC, Media, Pa) B)To gather visual acuity data for patients with known ocular problems, including cataract and maculopathy.

C)To correlate and compare the CVA visual acuity findings with the acuity measured with standard LogMAR acuity charts viewed under similar conditions of contrast and lighting

DETAILED DESCRIPTION:
The measurement of visual acuity involves the determination of the smallest high contrast target that can be resolved by the patient. Classically, this has been approached by the use of letter style optotypes, each having successively smaller stroke and gap resolution. More recently, the arrangements of letter charts have been redesigned with a logarithmic scale and with attention being paid to the uniformity of other effects such as crowding or of the choice of optotype. The resultant Ferris-Bailey-Lovie chart has become a standard for acuity testing, especially for clinical research. The letters of such acuity charts have a 0.1 logMAR step progression (1.26 X) between lines and have 5 letters per line. It has been noted that the logMAR chart could have greater resolution with finer steps between the lines and with improved repeatability by converting to a letter-by-letter scoring system.

While these advances have improved the resolution and reliability of acuity measures, they require relatively cumbersome wall charts and do not provide any of the advantages of an interactive program that would enable a threshold to be approached by stimulus presentation on both the seeing as well as non-seeing sides.

The Vimetrics CVA is an interactive computer device that measures threshold visual acuity by presenting a Landolt-C with the gap randomly tumbled in one of 4 positions to which the patient responds with a response pad. The threshold is approached in a logarithmic, staircase fashion to define the test subject's acuity threshold with a resolution similar to letter by letter scoring in chart testing but with the ability to rapidly test under a number of conditions of luminance and contrast that simulate activities of daily living.

The CVA determination of visual acuity under six conditions of contrast and lighting will be compared with that acquired by logMAR chart testing under similar conditions.

ELIGIBILITY:
General Exclusion Criteria:

those individuals whom the examiner determines cannot read the ETDRS letter chart to define vision and those individuals whom the examiner determines cannot respond to the computer presentation of the tumbled Landolt C by pressing one of the 4 buttons arranged in a diamond or by deflecting the joystick on the response pad held in the lap.

Normals:

Systemic Disease Exclusion Criteria: Persons with systemic disease that would interfere with vision will be excluded under the normal classification. Such diseases that would exclude a subject from this category would include diabetes, and other systemic diseases such as neurological disorders that the examiner determines may interfere with the vision of an eye.

Ocular Inclusion criteria:

For inclusion in the normal group an eye would have an ocular examination within three months that, in the least, included the following:

A visual acuity measured of 20/30 or better for which on examination the refractive error alone is determined to define the vision.

For individuals 65 years or greater, lens nuclear opalescence and brunescence that is less than or equal to NO3, NC3 according to the LOCS III grading system.

For individuals less than 65 years, lens nuclear opalescence and brunescence that is less than or equal to NO2, NC2, according to the LOCS III grading system.

Ocular Exclusion Criteria:

Media opacity or retinal or optic nerve pathology that the examiner determines would affect the measured vision.

For individuals aged 65 or greater, eyes with nuclear opalescence and brunescence, according to the LOCS III grading system greater than NO3, NC3 or with other opacities will be excluded.

Eyes with Cataracts:

General Inclusion Criteria:

Persons without systemic disease that would interfere with vision will be enrolled. Such diseases that would exclude a subject from this category would include diabetes, and other systemic diseases such as neurological disorders that the examiner determines may interfere with the vision of an eye.

Ocular Inclusion Criteria:

For inclusion an eye would have had an ocular examination within three months as per the stated protocol.

A visual acuity worse than 20/30. The determination on examination by the examiner that the lens opacity alone defines the vision. For individuals less than age 65 the nuclear cataract will be denser than NO2, NC2 or contain other components (posterior cortical or posterior sub capsular) that will be documented. For individuals 65 years of age or older, the nuclear cataract will be greater than NO3, NC3 or contain other components that define the vision.

Ocular Exclusion Criteria:

Eyes in which retinal or optic nerve pathology that the examiner determines would affect the measured vision.

Eyes with a best refracted chart acuity of 20/100 or worse because in such eyes the examiner will be prevented by the media opacity from adequately examining the fundus to determine if there is co-existent macular pathology.

Eyes with Maculopathy:

General Inclusion Criteria:

It is recognized that many individuals within this group will have diabetes or hypertension that may be the cause of the maculopathy or aggravate the maculopathy. However, such systemic diseases will not necessarily exclude such persons, unless the examiner determines that such diseases cause reduced vision in the eye that is not defined by the maculopathy.

Ocular Inclusion Criteria:

For inclusion an eye would have had an ocular examination within three months with components according to the protocol as stated.

A visual acuity with chart testing worse than 20/30 for which on examination the maculopathy alone is determined to define the vision.

Ocular Exclusion Criteria:

Eyes with a chart acuity of 20/400 or worse. Eyes having lens or optic nerve pathology that the examiner determines would affect the measured vision.

Eyes with dense cataract in which an adequate examination of the macula is prevented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Eye Clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Measurement of monocular Visual Acuity | Upon recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Sinclair, MD, Principal Investigator — Sinclair Technologies, LLC
Locations (2):
- Pennsylvania College of Optometry, Elkins Park, Pennsylvania, United States
- Gutstein Optik, Vienna, Austria

REFERENCES:
- [Background] Arditi A, Cagenello R. On the statistical reliability of letter-chart visual acuity measurements. Invest Ophthalmol Vis Sci. 1993 Jan;34(1):120-9. PMID 8425819
- [Background] Bourne RR, Rosser DA, Sukudom P, Dineen B, Laidlaw DA, Johnson GJ, Murdoch IE. Evaluating a new logMAR chart designed to improve visual acuity assessment in population-based surveys. Eye (Lond). 2003 Aug;17(6):754-8. doi: 10.1038/sj.eye.6700500. PMID 12928690
- [Background] Hazel CA, Elliott DB. The dependency of logMAR visual acuity measurements on chart design and scoring rule. Optom Vis Sci. 2002 Dec;79(12):788-92. doi: 10.1097/00006324-200212000-00011. PMID 12512687
- [Background] Raasch TW, Bailey IL, Bullimore MA. Repeatability of visual acuity measurement. Optom Vis Sci. 1998 May;75(5):342-8. doi: 10.1097/00006324-199805000-00024. PMID 9624699
- [Background] Bailey IL. New procedures for detecting early vision losses in the elderly. Optom Vis Sci. 1993 Apr;70(4):299-305. doi: 10.1097/00006324-199304000-00008. PMID 8502458
- [Background] Carkeet A. Modeling logMAR visual acuity scores: effects of termination rules and alternative forced-choice options. Optom Vis Sci. 2001 Jul;78(7):529-38. doi: 10.1097/00006324-200107000-00017. PMID 11503943